CLINICAL TRIAL: NCT01118299
Title: Amplatzer Cardiac Plug Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL00921
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Peripheral Thromboembolism
Keywords: ACP; Atrial Fibrillation; AF; A Fib; Stroke; Coumadin; Warfarin; Dabigatran; Pradaxa; Blood thinning medication; Left atrial appendage; LAA
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device (Experimental): AMPLATZER Cardiac Plug
  Interventions: Device: AMPLATZER Cardiac Plug
- Optimal Medical Therapy (control) (Active Comparator): Warfarin Dabigatran
  Interventions: Device: AMPLATZER Cardiac Plug

INTERVENTIONS:
Device: AMPLATZER Cardiac Plug — AMPLATZER Cardiac Plug is a percutaneous transcatheter device

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the ACP in subjects with nonvalvular atrial fibrillation by demonstrating that the device is non-inferior to optimal medical therapy (OMT) with respect to the primary effectiveness endpoint and superior to OMT with respect to primary safety endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a documented history of paroxysmal, persistent or permanent nonvalvular atrial fibrillation
* Subject must be ≥18 years of age
* Subject must be on warfarin or dabigatran therapy
* Subject must be eligible for long term warfarin or dabigatran therapy
* Subject must have a CHADS(2) score of 2 or greater

Summary of Exclusion Criteria:

* Subject who requires warfarin or dabigatran for a condition other than AF
* Subject who is on clopidogrel or another P2Y12 platelet inhibitor such as prasugrel or ticagrelor
* Subject who has an absolute or relative contraindication to aspirin, or warfarin and dabigatran
* Subject with a New York Heart Association (NYHA) classification equal to IV
* Subject with an implanted or surgical repair atrial septal defect (ASD) device or patent foramen ovale (PFO) device
* Subject with aortic or mitral valve regurgitation of grade 2+ or greater
* Subject with left ventricular ejection fraction (LVEF) ≤30
* Subject with mitral or aortic prosthetic valve
* Subject with a history of hemorrhagic or aneurysmal stroke
* Subject with a history of previous radio frequency (RF) ablation for atrial fibrillation
* Subject with a body mass index (BMI) ≥40
* Subject with a history of acute or recent MI, or unstable angina, or coronary artery bypass graft surgery (within 6 months)
* Subject who is on aspirin dose therapy greater than 81mg/day at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-04-26 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Good Samaritan Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - South Denver Cardiology Associates, Littleton, Colorado
  - Emory Midtown Hospital and Emory University Hospital, Atlanta, Georgia
  - St. Joseph's Hospital and Research Institute, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Providence Hospital, Southfield, Michigan
  - St. Cloud Hospital/CentraCare Heart and Vascular Clinic, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roper Hospital/PMG Research of Charleston, Charleston, South Carolina
  - Memorial Hermann Hospital, Houston, Texas
  - Aspirus Heart & Vascular Institute, Wausau, Wisconsin

REFERENCES:
- See also: What is Atrial Fibrillation - Fact Sheet — http://www.americanheart.org/downloadable/heart/119618028569709%20WhatisAtrialFibrillation%209_07.pdf
- See also: Overview of Atrial Fibrillation — http://www.nhlbi.nih.gov/health/dci/Diseases/af/af_what.html
- See also: Let's Talk about Stroke, TIA and Warning Signs - Fact Sheet — http://www.americanheart.org/downloadable/heartsmart/118582358042250-0066%20ASA%20TIAWrngSigns_4-07.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device | Optimal Medical Therapy (Control)
Started | 68 | 29
Completed | 45 | 0
Not Completed | 23 | 29
Not completed — Death | 7 | 5
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Enrollment Closure, Protocol Amendment | 6 | 15

BASELINE CHARACTERISTICS:
Population: All 97 randomized subjects were part of the baseline population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Device | Optimal Medical Therapy (Control) | Total
Number analyzed (Participants) | 68 | 29 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.0 (8.5) | 73.4 (10.0) | 73.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 45 | 18 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
CHADS2 Score [Count of Participants; unit: Participants] — CHADS2 (Congestive heart failure, Hypertension, Age, Diabetes, Stroke or TIA )score can help doctor figure out how likely patient will have a stroke and decide if patient needs to take something to help prevent one. our score will be between 0 and 6 points:
  Zero: You aren't likely to have a stroke.
  One point: You have a medium risk of stroke.
  Two or more points: Your odds of having a stroke are medium to high, and your doctor probably will prescribe a blood thinner. You may hear your doctor use the medical term for that kind of medicine: oral anticoagulant.
  Participants
    Chads2 Score 0 | 0 | 0 | 0
    Chads2 Score 1 | 0 | 0 | 0
    Chads2 Score 2 | 38 | 17 | 55
    Chads2 Score 3 | 20 | 7 | 27
    Chads2 Score 4 | 7 | 4 | 11
    Chads2 Score 5 | 2 | 1 | 3
    Chads2 Score 6 | 1 | 0 | 1
History of Atrial Fibrillation [Count of Participants; unit: Participants]
  Paroxysmal | 32 | 19 | 51
  Persistent | 21 | 7 | 28
  Permanent | 15 | 3 | 18
Rhythm Status at Baseline [Count of Participants; unit: Participants] — Population: One subject did not have a baseline ECG performed. Hence the denominator is for 96 subjects.
  Participants
    number analyzed (Participants) | 67 | 29 | 96
    Paced Rhythm | 17 | 15 | 32
    Atrial Fibrillation | 29 | 5 | 34
    Sinus Rhythm | 19 | 7 | 26
    Other Arrhythmias or Conduction Disturbance | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Acute Safety - Procedure Related SAEs From Randomization Through Discharge For Device Arm Only
Description: An analysis comparing the rate of procedure related serious adverse events that occur in the device arm to a performance goal determined from literature reported rates for similar procedural techniques.
  The study as designed was intended to determine the difference in efficacy and safety between the device and control arm (subjects treated with OMT).
  However, due to early enrollment closure, the three primary endpoints were not analyzed as specified in the original trial protocol. As the Control arm subjects exited the study early, no sufficient data was available to summarize any endpoints. The three primary endpoints as mentioned in the Appendix D of the clinical investigational plan (Revision 06, dated September 2014) were summarized for the Device arm below. The secondary endpoint analysis requirement was removed from the protocol.
Time Frame: From Randomization to Discharge Visit
Population: No data were collected for the Control Arm/Group due to early enrollment closure and the pre-specified analysis was revised accordingly to report data for only the Device Arm.
Measure: Number; unit: events
Groups:
- Device Arm: Subjects who received the ACP device
Arm/Group | Device Arm
Number analyzed (Participants) | 68
events
  Device Embolization | 3
  Pleural Effusion | 1
  Hematoma | 1
  Pericardial Tamponade | 3
  Cardiac Perforation* | 1
  Pericardial Effusion | 1
  Cardiogenic Shock* | 1
  Pericarditis* | 1

2. Primary Outcome: Long-term Safety - Device Arm Only
Description: All-Cause Mortality and Major Bleeds Through 2 years in device arm subjects only. The study as designed was intended to determine the difference in efficacy and safety between the device and control arm (subjects treated with OMT).
  However, due to early enrollment closure, the three primary endpoints were not analyzed as specified in the original trial protocol. As the Control arm subjects exited the study early, no sufficient data was available to summarize any endpoints. The three primary endpoints as mentioned in the Appendix D of the clinical investigational plan (Revision 06, dated September 2014) were summarized for the Device arm. The secondary endpoint analysis requirement was removed from the protocol.
Time Frame: Randomization to 2 year follow-up
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Device Arm
Number analyzed (Participants) | 68
Events
  Empyema (Major Bleeding) | 1
  Hemothorax (Major Bleeding) | 1
  Hematoma (Major Bleeidng) | 1
  Bleeding (Major Bleeding) | 1
  Respiratory Failure (Death) | 2
  Congestive Heart Failure (Death) | 1
  Device Embolization (Death) | 1

3. Primary Outcome: Effectiveness Endpoint - Device Arm Only
Description: Occurrence of ischemic stroke and peripheral thromboembolism in the device arm. The study as designed was intended to determine the difference in efficacy and safety between the device and control arm (subjects treated with OMT).
  However, due to early enrollment closure, the three primary endpoints were not analyzed as specified in the original trial protocol. As the Control arm subjects exited the study early, no sufficient data was available to summarize any endpoints. The three primary endpoints as mentioned in the Appendix D of the clinical investigational plan (Revision 06, dated September 2014) were summarized for the Device arm. The secondary endpoint analysis requirement was removed from the protocol.
Time Frame: Randomization through 2 year follow up
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Device Arm
Number analyzed (Participants) | 68
events
  Ischemic Stroke | 2
  Peripheral Thromboembolism | 0

ADVERSE EVENTS:
Time Frame: 5 Years
Description: Abbott's internal AE coding system used for these AEs. All AEs coded as Cardiac Disorders.
Arm/Group | Device | Optimal Medical Therapy (Control)
All-Cause Mortality (participants affected / at risk) | 7/68 | 5/29
Serious Adverse Events (participants affected / at risk) | 52/68 | 15/29
Other Adverse Events (participants affected / at risk) | 61/68 | 15/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=68) | Optimal Medical Therapy (Control) (N=29)
Abnormal Coagulation Parameter (Cardiac disorders) | 1 (1) | 1 (1)
Abnormal Lab Value (Cardiac disorders) | 1 (1) | 0 (0)
Acute Bronchitis (Cardiac disorders) | 2 (2) | 1 (1)
Acute Erosive Gastritis (Cardiac disorders) | 1 (1) | 0 (0)
Acute Pancreatitis (Cardiac disorders) | 2 (3) | 0 (0)
Acute Renal Failure (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arthritis (Cardiac disorders) | 1 (1) | 0 (0)
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 8 (10) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Bacteremia (Cardiac disorders) | 1 (1) | 1 (1)
Bacterial Infections (Cardiac disorders) | 3 (3) | 0 (0)
Benign Tumors (Cardiac disorders) | 1 (1) | 0 (0)
Bleeding (Cardiac disorders) | 1 (1) | 0 (0)
Breast Cancer (Cardiac disorders) | 0 (0) | 1 (1)
Cancer (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Perforation* (Cardiac disorders) | 1 (1) | 0 (0) — * This event was considered as sub-event of the master event for Pericardial Tamponade.
Cardiogenic Shock* (Cardiac disorders) | 1 (1) | 0 (0) — * This event was considered as sub-event of the master event for Pericardial Tamponade.
Cellulitis (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral Aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cervical Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 4 (4) | 0 (0)
Cholecystitis (Cardiac disorders) | 2 (2) | 0 (0)
Chronic Obstructive Pulmonary Disease (COPD) (Cardiac disorders) | 2 (6) | 1 (1)
Closed Head Injury (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Cardiac disorders) | 1 (1) | 0 (0)
Confusion (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 5 (6) | 6 (7)
Constrictive Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Deep Vein/Venous Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Cardiac disorders) | 1 (1) | 0 (0)
Delirium (Cardiac disorders) | 1 (1) | 0 (0)
Device Closure of ASD (Cardiac disorders) | 1 (1) | 0 (0)
Device Embolization (Cardiac disorders) | 4 (4) | 0 (0)
Drug Side Effect (Cardiac disorders) | 0 (0) | 1 (2)
Dysphagia (Cardiac disorders) | 2 (2) | 0 (0)
Dyspnea (Cardiac disorders) | 0 (0) | 1 (1)
Ear Infection (Cardiac disorders) | 1 (1) | 0 (0)
Elective Procedure (Cardiac disorders) | 0 (0) | 1 (1)
Elective Surgery (Cardiac disorders) | 1 (1) | 2 (2)
Emphysema (Cardiac disorders) | 0 (0) | 1 (1)
Empyema (Cardiac disorders) | 1 (1) | 0 (0)
Encephalopathy (Cardiac disorders) | 1 (1) | 0 (0)
Esophageal Laceration and Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Cardiac disorders) | 1 (1) | 0 (0)
Fracture (Cardiac disorders) | 1 (1) | 0 (0)
Gout (Cardiac disorders) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Hemarthrosis (Cardiac disorders) | 1 (2) | 0 (0)
Hematoma (Cardiac disorders) | 2 (2) | 1 (1)
Hemorrhagic Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Hemothorax (Cardiac disorders) | 1 (1) | 0 (0)
Hip Fracture (Cardiac disorders) | 1 (1) | 1 (1)
Hydrocephalus (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive Crisis (Cardiac disorders) | 1 (1) | 0 (0)
Hyponatremia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Ischemic Stroke (Cardiac disorders) | 2 (2) | 2 (2)
Knee Pain (Cardiac disorders) | 1 (1) | 0 (0)
Low Back Pain (Cardiac disorders) | 1 (1) | 0 (0)
Lumbar Disc Displacement (Cardiac disorders) | 0 (0) | 1 (1)
Lumbar Spondylosis (Cardiac disorders) | 1 (1) | 0 (0)
Melena (Cardiac disorders) | 1 (1) | 0 (0)
Migraine (Cardiac disorders) | 1 (1) | 0 (0)
Mononucleosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Osteoarthritis/Degenerative Joint Disease (Cardiac disorders) | 2 (3) | 0 (0)
Other: Pancreatic pseudocyst (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 5 (5) | 0 (0)
Pericardial Tamponade (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis* (Cardiac disorders) | 2 (3) | 0 (0) — * This event was considered as sub-event of the master event for Pericardial Tamponade.
Peripheral Arterial Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Persistent Atrial Fibrillation (Cardiac disorders) | 3 (6) | 0 (0)
Pleural Effusion (Cardiac disorders) | 3 (3) | 0 (0)
Pneumonia (Cardiac disorders) | 4 (8) | 2 (2)
Polyneuropathy (Cardiac disorders) | 1 (1) | 0 (0)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Cardiac disorders) | 1 (1) | 0 (0)
Renal Failure (Cardiac disorders) | 1 (1) | 0 (0)
Renal Insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Respiratory Failure (Cardiac disorders) | 3 (4) | 0 (0)
Sepsis (Cardiac disorders) | 3 (5) | 2 (2)
Sick Sinus Syndrome (Cardiac disorders) | 2 (2) | 1 (1)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 2 (2) | 2 (2)
Sinusitis (Cardiac disorders) | 1 (1) | 0 (0)
Spells (Cardiac disorders) | 2 (2) | 0 (0)
Spinal Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 1 (1)
Transient Ischemic Attack (TIA) (Cardiac disorders) | 0 (0) | 1 (1)
Trauma (Cardiac disorders) | 1 (1) | 0 (0)
Unstable Angina (Cardiac disorders) | 1 (2) | 0 (0)
VASC Bleeding (Cardiac disorders) | 2 (2) | 0 (0)
VASC Hematoma (Cardiac disorders) | 3 (3) | 0 (0)
Vancomycin-Resistant Enterococcus (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Viral Gastroenteritis (Cardiac disorders) | 1 (1) | 0 (0)
Visual Disturbance (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=68) | Optimal Medical Therapy (Control) (N=29)
Abdominal Bloating (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Cardiac disorders) | 1 (1) | 1 (1)
Abnormal Coagulation Parameter (Cardiac disorders) | 1 (2) | 1 (1)
Abnormal Lab Value (Cardiac disorders) | 3 (3) | 0 (0)
Abnormal Renal Function (Cardiac disorders) | 1 (1) | 0 (0)
Abrasion (Cardiac disorders) | 2 (3) | 0 (0)
Acute Bronchitis (Cardiac disorders) | 4 (4) | 1 (1)
Acute Kidney Injury (Cardiac disorders) | 1 (1) | 0 (0)
Acute Renal Failure (Cardiac disorders) | 0 (0) | 2 (2)
Air Embolus (Cardiac disorders) | 1 (1) | 0 (0)
Allergic Drug Reaction (Cardiac disorders) | 1 (1) | 0 (0)
Allergy (Cardiac disorders) | 1 (1) | 0 (0)
Anemias (Cardiac disorders) | 1 (1) | 1 (1)
Animal Bite (Cardiac disorders) | 0 (0) | 1 (1)
Anxiety (Cardiac disorders) | 1 (1) | 0 (0)
Anxiety Reaction (Cardiac disorders) | 1 (1) | 0 (0)
Aortic Aneurysms (Cardiac disorders) | 0 (0) | 2 (2)
Aortic Valve Stranding (Cardiac disorders) | 1 (1) | 0 (0)
Aphasia (Cardiac disorders) | 0 (0) | 1 (1)
Arm Fracture (Cardiac disorders) | 2 (2) | 0 (0)
Arterial Hypertension/Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Arthritis (Cardiac disorders) | 1 (1) | 1 (1)
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (Cardiac disorders) | 1 (1) | 0 (0)
Asthma (Cardiac disorders) | 1 (1) | 0 (0)
Asymptomatic Ischemic Stroke (Cardiac disorders) | 3 (3) | 0 (0)
Atelectasis (Cardiac disorders) | 3 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 6 (9) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 2 (2)
Back Pain (Cardiac disorders) | 2 (2) | 1 (1)
Bee Sting (Cardiac disorders) | 1 (1) | 0 (0)
Behavior Alterations (Cardiac disorders) | 0 (0) | 1 (1)
Bells Palsy (Cardiac disorders) | 0 (0) | 1 (1)
Bleeding (Cardiac disorders) | 5 (5) | 0 (0)
Bronchitis (Cardiac disorders) | 2 (2) | 0 (0)
Bruise/Purpura Simplex (Cardiac disorders) | 5 (6) | 1 (1)
Bursitis (Cardiac disorders) | 1 (1) | 0 (0)
Carpal Tunnel (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Cardiac disorders) | 1 (1) | 1 (1)
Cellulitis (Cardiac disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 3 (3) | 2 (3)
Chronic Obstructive Pulmonary Disease (COPD) (Cardiac disorders) | 3 (3) | 0 (0)
Chronic Renal Failure (Cardiac disorders) | 1 (1) | 0 (0)
Chronic Subdural Hematoma (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Cardiac disorders) | 1 (1) | 0 (0)
Colon Polyps (Cardiac disorders) | 0 (0) | 1 (1)
Common Cold/Upper Respiratory Tract Infection (Cardiac disorders) | 4 (4) | 0 (0)
Compressive Effect On Nerve (Cardiac disorders) | 1 (1) | 0 (0)
Concussion (Cardiac disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Cardiac disorders) | 0 (0) | 1 (1)
Contusion (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Cardiac disorders) | 1 (1) | 0 (0)
Decreased Appetite (Cardiac disorders) | 1 (1) | 0 (0)
Decreased Sphincter Tone (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Cardiac disorders) | 1 (2) | 0 (0)
Depression (Cardiac disorders) | 3 (3) | 1 (1)
Device Malposition or Malfunction (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhea (Cardiac disorders) | 1 (1) | 1 (1)
Diastolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Difficulty Catching Breath (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia/Double Vision (Cardiac disorders) | 1 (1) | 0 (0)
Diverticulitis (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Cardiac disorders) | 3 (4) | 0 (0)
Drug Rash (Cardiac disorders) | 1 (1) | 0 (0)
Drug Side Effect (Cardiac disorders) | 2 (3) | 1 (1)
Dyspepsia (Cardiac disorders) | 2 (2) | 1 (1)
Dysphagia (Cardiac disorders) | 3 (3) | 0 (0)
Dyspnea (Cardiac disorders) | 7 (7) | 1 (1)
Earache (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 9 (9) | 2 (2)
Elective Procedure (Cardiac disorders) | 0 (0) | 1 (1)
Elective Surgery (Cardiac disorders) | 1 (1) | 0 (0)
Emesis/Vomiting (Cardiac disorders) | 0 (0) | 1 (1)
Encephalopathy (Cardiac disorders) | 1 (1) | 0 (0)
Epididymitis (Cardiac disorders) | 1 (1) | 0 (0)
Epistaxis (Cardiac disorders) | 2 (2) | 2 (2)
Erectile Dysfunction Symptoms (Cardiac disorders) | 1 (1) | 0 (0)
Eye Swelling (Cardiac disorders) | 0 (0) | 1 (1)
Fall (Cardiac disorders) | 6 (7) | 2 (2)
Fatigue/Generalized Fatigue (Cardiac disorders) | 3 (3) | 0 (0)
Fever (Cardiac disorders) | 1 (1) | 0 (0)
Folliculitis (Cardiac disorders) | 0 (0) | 1 (1)
Fracture (Cardiac disorders) | 2 (2) | 1 (1)
Fungal Skin Infection (Cardiac disorders) | 1 (1) | 1 (1)
Gastritis (Cardiac disorders) | 2 (2) | 0 (0)
Gastrointestinal Bleeding (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal Illness (Cardiac disorders) | 1 (1) | 0 (0)
Gingival Bleeding (Cardiac disorders) | 0 (0) | 1 (1)
Gout (Cardiac disorders) | 1 (1) | 0 (0)
Headache (Cardiac disorders) | 1 (1) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Heartburn (Cardiac disorders) | 0 (0) | 1 (1)
Hemarthrosis (Cardiac disorders) | 0 (0) | 1 (1)
Hematoma (Cardiac disorders) | 2 (2) | 0 (0)
Hematuria (Cardiac disorders) | 2 (3) | 0 (0)
Hemoptysis (Cardiac disorders) | 1 (1) | 0 (0)
Hepatic and Biliary Disorders (Cardiac disorders) | 1 (1) | 0 (0)
Hip Pain (Cardiac disorders) | 2 (2) | 0 (0)
Hyperkalemia (Cardiac disorders) | 2 (2) | 0 (0)
Hypernatremia (Cardiac disorders) | 1 (1) | 0 (0)
Hypokalemia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 8 (8) | 0 (0)
Hypoxemia (Cardiac disorders) | 1 (1) | 1 (1)
Incidental Finding of Stroke (Cardiac disorders) | 1 (1) | 0 (0)
Intracerebral Haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Iron-Deficiency Anemia (Cardiac disorders) | 1 (1) | 0 (0)
Junctional Escape Rhythm/Intermittent Junctional Rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Knee Pain (Cardiac disorders) | 1 (1) | 1 (1)
Lacerations (Cardiac disorders) | 1 (1) | 1 (1)
Lightheadedness (Cardiac disorders) | 1 (1) | 0 (0)
Low Back Pain (Cardiac disorders) | 2 (2) | 0 (0)
Lung Crackles (Cardiac disorders) | 1 (1) | 0 (0)
Memory Difficulty (Cardiac disorders) | 1 (1) | 0 (0)
Microhemorrhage (Cardiac disorders) | 2 (2) | 0 (0)
Mitral Valve Regurgitation/Mitral Insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Cardiac disorders) | 1 (1) | 2 (2)
Nausea (Cardiac disorders) | 2 (2) | 0 (0)
Neck Pain (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Cardiac disorders) | 1 (1) | 0 (0)
Nocturia (Cardiac disorders) | 1 (1) | 0 (0)
Non-Specific EKG Change (Cardiac disorders) | 1 (1) | 0 (0)
Numbness (Cardiac disorders) | 5 (5) | 0 (0)
Onychomycosis (Cardiac disorders) | 0 (0) | 1 (1)
Overhydration (Cardiac disorders) | 1 (1) | 0 (0)
Pain (Cardiac disorders) | 3 (4) | 1 (1)
Palpitations (Cardiac disorders) | 5 (5) | 2 (2)
Parkinson's Disease (Cardiac disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 5 (5) | 0 (0)
Peripheral Venous Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Persistent Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Phlebitis (Cardiac disorders) | 1 (1) | 0 (0)
Plantar Fasciitis (Cardiac disorders) | 1 (1) | 0 (0)
Pleural Effusion (Cardiac disorders) | 2 (4) | 1 (1)
Pleuretic Pain (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Cardiac disorders) | 3 (4) | 3 (3)
Pneumothorax (Cardiac disorders) | 1 (1) | 0 (0)
Post-Menopausal Bleeding (Cardiac disorders) | 1 (1) | 0 (0)
Pressure Sores (Cardiac disorders) | 0 (0) | 2 (2)
Psychogenic Event (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Ramsay Hunt Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Rash (Cardiac disorders) | 1 (1) | 1 (1)
Residual Interatrial Communication (Cardiac disorders) | 7 (7) | 0 (0)
Respiratory Illness (Cardiac disorders) | 1 (1) | 0 (0)
Rhinitis (Cardiac disorders) | 1 (1) | 0 (0)
ST Segment Changes (Cardiac disorders) | 2 (2) | 0 (0)
Sciatica (Cardiac disorders) | 1 (1) | 0 (0)
Shingles (Cardiac disorders) | 4 (4) | 0 (0)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 2 (2) | 0 (0)
Sinusitis (Cardiac disorders) | 2 (3) | 0 (0)
Skin Cancer (Cardiac disorders) | 1 (1) | 0 (0)
Skin Lesions (Cardiac disorders) | 1 (1) | 1 (1)
Skin Ulcer (Cardiac disorders) | 1 (1) | 0 (0)
Sore Throat (Cardiac disorders) | 5 (6) | 0 (0)
Spells (Cardiac disorders) | 1 (3) | 2 (2)
Stupor (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Temporomandibular Joint (Cardiac disorders) | 1 (1) | 0 (0)
Tendosynovitis (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombus on Device (Cardiac disorders) | 2 (2) | 0 (0)
Thyroid Disorders (Cardiac disorders) | 2 (2) | 0 (0)
Toe Inflammation (Cardiac disorders) | 1 (1) | 0 (0)
Transient Imbalance (Cardiac disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (TIA) (Cardiac disorders) | 0 (0) | 1 (2)
Trauma (Cardiac disorders) | 1 (1) | 1 (1)
Tremor (Cardiac disorders) | 1 (1) | 1 (1)
Uncontrolled Blood Sugar (Cardiac disorders) | 1 (1) | 0 (0)
Unsustained/Nonsustained Ventricular Tachy/Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) — Unsustained/Nonsustained Ventricular Tachy/Cardiac Arrhythmia: Other - Non-sustained runs of VT, Ventricular Ectopic Beats/Premature Ventricular Contractions/Premature Ventricular Beats
Urinary Incontinence (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Retention (Cardiac disorders) | 3 (3) | 1 (1)
Urinary Tract Infections (Cardiac disorders) | 6 (7) | 1 (1)
VASC Bleeding (Cardiac disorders) | 10 (10) | 0 (0)
VASC Bruise (Cardiac disorders) | 3 (3) | 0 (0)
VASC Hematoma (Cardiac disorders) | 7 (7) | 0 (0)
VASC Pseudoaneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Cardiac disorders) | 2 (2) | 0 (0)
Visual Disturbance (Cardiac disorders) | 1 (1) | 1 (1)
Weakness (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/99/NCT01118299/Prot_SAP_000.pdf